CLINICAL TRIAL: NCT03229200
Title: Extended Treatment Protocol for Subjects Continuing to Benefit From Ibrutinib After Completion of Ibrutinib Clinical Trials.
Brief Title: Extended Treatment Protocol for Subjects Continuing to Benefit From Ibrutinib.
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Pharmacyclics Switzerland GmbH (Industry)
Collaborators: Janssen Biotech, Inc., including Johnson & Johnson (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1145-LT; 2016-004356-30 (EudraCT Number)
Record Dates: First submitted 2017-06-05; First posted 2017-07-25 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Leukemia, B-cell; Graft Vs Host Disease; Solid Tumor
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Leukemia, B-Cell; Graft vs Host Disease | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ibrutinib (Experimental): Treatment with Ibrutinib, once daily until disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Subjects will continue with the current ibrutinib dosing regimen established in the parent ibrutinib study.

SUMMARY:
Multicenter, open-label, prospective treatment protocol that provides continued access to ibrutinib to subjects who have completed parent ibrutinib studies, are still benefitting from treatment with ibrutinib, and have no access to commercial ibrutinib for their underlying disease within their region.

DETAILED DESCRIPTION:
Multicenter, open-label, prospective treatment protocol that provides continued access to ibrutinib to subjects who have completed parent ibrutinib studies, are still benefitting from treatment with ibrutinib, and have no access to commercial ibrutinib for their underlying disease within their region.

Subjects enrolled in this treatment protocol will receive oral continuous dosing with ibrutinib at the same dose and schedule they were receiving at the end of the respective parent study. Treatment may be continued as long as the subjects continue to derive benefit from treatment with ibrutinib until such time that ibrutinib becomes commercially available for the indication of the parent study.

Clinical evaluations (including safety assessments) will be performed per local standard of care for each disease that was studied in the parent protocol. At each visit, all ongoing and new onset non-serious AEs leading to dose reduction or discontinuation, serious adverse events (SAEs), adverse events of special interest (AESI), pregnancy events, other malignancies, and special reporting situations will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have participated in an eligible ibrutinib clinical trial, may derive clinical benefit from continued treatment or restart of treatment with ibrutinib in the opinion of the treating physician and does not have access to commercial ibrutinib within their region and/or the drug is not reasonably accessible to the patient within the respective region.
* Ongoing continuous treatment with ibrutinib.
* Subject must have completed all assessments in their parent protocol and want to continue treatment with ibrutinib.
* Subject or their legally authorized representative must voluntarily sign and date an informed consent approved by an independent ethics committee (IEC)/institutional review board (IRB) to the long term treatment extension protocol and not withdrawn consent from the parent study.
* Male and female subjects of reproductive potential who agree to use both a highly effective method of birth control and a barrier method during the period of therapy and for 90 days after the last dose of drug.

Exclusion Criteria:

* Meeting any requirement in the parent protocol to permanently discontinue ibrutinib treatment.
* Any condition or situation which, in the opinion of the treating physician, may interfere significantly with a subject's participation in the protocol.
* Female subjects who are pregnant, or breastfeeding, or planning to become pregnant while enrolled in this protocol or within 90 days of last dose of drug treatment. Male subjects who plan to father a child while enrolled in this protocol or within 90 days after the last dose of drug treatment.
* Unwilling or unable to participate in all required evaluations and procedures.
* Unable to understand the purpose and risks of the protocol and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2027-05-10 (Estimated); Study Completion 2027-05-10 (Estimated)

PRIMARY OUTCOMES:
Characterize the drug safety profile by collecting long-term safety data for ibrutinib. | Up to 3 years and will be re-evaluated on an ongoing basis.
  Number of participants with treatment emergent serious adverse events and adverse events of special interest as assessed by CTCAE v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Wu, Study Director — AbbVie
Locations (98):
- United States (34):
  - Providence Health System - Southern California d/b/a Roy and Patricia Disney Family Cancer Center, The Roy & Patricia Disney Family Cancer Center, Burbank, California
  - City Of Hope National Medical Center, Duarte, California
  - UCSD Moores Cancer Center, La Jolla, California
  - University of California Los Angeles (UCLA), Los Angeles, California
  - Stanford University, Stanford, California
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Norton Medical Plaza II, 3991 Dutchmans Lane, Louisville, Kentucky
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - TRIO - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - John Theurer Cancer Center, Hackensack UMC, Hackensack, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Northwell Health, New Hyde Park, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Mid Ohio Oncology/Hematology Inc., DBA The Mark H. Zangmeister Center, Columbus, Ohio
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - M.D. Anderson Cancer Centre, Houston, Texas
  - US Oncology Research, LLC, The Woodlands, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Swedish Cancer Institute, Seattle, Washington
  - Northwest Cancer Specialists, Compass Oncology, Vancouver, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
- Australia (9):
  - St. George Hospital, Kogarah, New South Wales
  - Concord Repatriation General Hospital - Haematology Clinical Trials, Sydney, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Ballarat Health Services, Ballarat, Victoria
  - Eastern Health, Box Hill, Victoria
  - Monash Health-Monash Medical Centre, Clayton, Victoria
  - St Vincent Hospital, Fitzroy, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Canada (3):
  - QEII Health Science Centre, Halifax, Nova Scotia
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec
- Czechia (5):
  - University Hospital Hradec Kralove, Hradec Králové, Královéhradecký kraj
  - Hematology and Oncology Masaryk University Hospital Brno, Brno
  - University Hospital Pilsen, Pilsen
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Charles University Hospital, Prague, Prague
- France (3):
  - CHU Hotel Dieu, Nantes, Loire Atlantique
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier Saint Brieuc, Saint-Brieuc
- Central Hospital of Southern Pest - National Institute of Hematology and Infectious Diseases, Dept of Hematology and Stem Cell, Budapest, Hungary
- Italy (7):
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele IRCCS, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia
  - Azienda Ospedaliera CittÃ della Salute e della Scienza di Torino, Torino
  - Azienda Sanitaria Universitaria Integrata Udine, Udine
- New Zealand (2):
  - Middlemore Hospital, Papatoetoe, Auckland
  - North Shore Hospital, Auckland
- Poland (4):
  - Szpital Specjalistyczny w Brzozowie, Oddział Hematologii Onkologicznej z Klinicznym Oddziałem Przeszczepiania Szpiku, Brzozów, Podkarpackie Voivodeship
  - Klinika Hematologii i Transplantologii, Gdansk, Pomeranian Voivodeship
  - SPZOZ ZSM w Chorzowie, Chorzów, Silesian Voivodeship
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika, Lodz
- Russia (5):
  - Nizhniy Novgorod Regional Clinical Hospital n.a. N.A. Semashko, Nizhny Novgorod, Nizhegorodskaya
  - SBI of Ryazan region "Regional Clinical Hospital", Ryazan, Ryazan Oblast
  - Russian Scientific and Research Institute of Hematology and Transfusiology of Federal Medical Biological Agency, Saint Petersburg
  - Almazov National Medical Research Centre, Saint Petersburg
  - Yaroslavl Regional Clinical Hospital, Yaroslavl
- Kyungpook National University Hospital (KNUH), Daegu, South Korea
- Spain (7):
  - ICO - Hospital Germans Trias I Pujol, Badalona, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Vall d'Hebron, Barcelona
  - Hospital de Sanata Creus i Sant Pau, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - University Hospital of Salamanca, Salamanca
- Sweden (3):
  - Sunderby hospital, Luleå, Norrbotten County
  - Södra Älvsborg Hospital Borås, Borås
  - Karolinska Universitetssjukhuset, Solna, Solna
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (5):
  - Pamukkale University Medical Faculty, Denizli, Pamukkale
  - Ankara Universitesi Tip Fakultesi Hastanesi, Ankara
  - Gazi University, Ankara
  - VKV American Hospital, Istanbul
  - Dokuz Eylul University, Izmir
- Ukraine (3):
  - CNE CCOHTPC of Cherkasy Regional Council, Cherkasy
  - CNCE City Clinical Hospital 4 of Dnipro City Council, Dnipro
  - SI Institute of Blood Pathology and Transfusion Medicine of AMSU, Lviv
- United Kingdom (4):
  - University Hospital of Wales, Cardiff
  - Leeds Teaching Hospitals NHS, Leeds
  - University College Hospitals NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No